CLINICAL TRIAL: NCT03804255
Title: Biomarker Testing in Common Solid Cancers: An Assessment of Current Practices in Precision Oncology in the Community Setting
Brief Title: Assessment of Current Biomarker Testing Practices for Common Solid Cancers in Precision Oncology in the Community Setting
Status: Withdrawn | Type: Observational
Why Stopped: Study closed before patients enrolled
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: EAQ161CD; NCI-2018-01707 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ161CD (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ161CD (Other: DCP); EAQ161CD (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma; Community Practice; Lung Carcinoma; Melanoma; Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (survey): Participants complete a self-administered web-based Biomarker Survey and may also complete an Outcome Validation Survey.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete surveys

SUMMARY:
This trial assesses current biomarker testing practices for common solid cancers in precision oncology in the community setting. Cancer biomarkers are used for diagnosing the disease, determining prognosis, predicting response to a targeted therapy, or monitoring response to therapy. Testing quality, including accuracy and timeliness, is imperative for correct disease prognosis and identification of patients who may or may not benefit from a targeted therapy. Assessing current biomarker testing practices may help doctors identify gaps and variations in testing as well as on potential ?best practices? that may be informative and generalizable to community oncology programs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine capacity of pathology practices within National Cancer Institute (NCI) Community Oncology Research Program (NCORP) components/subcomponents for testing guideline-recommended biomarkers, including whether these biomarkers are tested, and how, i.e. what technologies are used and what ordering and testing processes / protocols have been implemented.

II. Determine capacity for testing for novel biomarkers and tumor molecular profiling, i.e. whether these biomarkers are tested and how, i.e. what technologies are used what ordering and testing processes/protocols have been implemented.

III. For findings in Objectives 1 and 2, determine factors influencing the heterogeneity of capacity for biomarker testing, particularly those factors that are modifiable (based on the conceptual framework above), such as cost, complexity, technologic complexity, lack of familiarity, physician and patient demand.

OUTLINE:

Participants complete a self-administered web-based Biomarker Survey and may also complete an Outcome Validation Survey.

ELIGIBILITY:
Inclusion Criteria:

* The study population is all onsite pathology practices within NCORP components and subcomponents that provide services to adult oncology groups.
* An onsite pathology practice is a laboratory (lab) that is financially administered and operated by an NCORP component or subcomponent. This excludes commercial reference laboratories, such as Quest and LabCorp. To describe biomarker testing practices across NCORP components/subcomponents, we will use the pathology practice as the unit of analysis. Participating components/subcomponents should meet [element A] AND [at least one element of B OR C OR D] AND element E.

  * A) NCORP component/subcomponent provides services to adult oncology groups.
  * B) A single onsite pathology lab (and its set of testing practices), may provide biomarker/pathology testing services to one or more components or subcomponents. Irrespective of the number of components/subcomponents that use this pathology lab, we will consider this as one pathology practice, and one unit of analysis.
  * C) Several onsite pathology labs may provide services to one NCORP component or subcomponent, e.g. if the NCORP component or subcomponent represents a health system with several hospitals, and each hospital may have its own onsite pathology lab, with each pathology lab following its own set of testing practices. Therefore, each lab will represent one pathology practice and one unit of analysis.
  * D) More than one onsite pathology lab may use a common set of testing practices and provide services to one or more NCORP components or subcomponents. Given common testing practices, we will consider these labs as one pathology practice, and one unit of analysis.
  * E) The pathology practice has an informed individual who is willing to serve as a representative and gather information to complete the assessment items. This person typically is the pathology practice medical director, pathology practice administrative director and/or their designees.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Onsite pathology practices within NCORP components and subcomponents that provide services to adult oncology groups
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Presence of reflexive testing protocols for guideline-recommended biomarkers | Up to 9 months
  Defined as standing protocols that do not require an oncologist order for each of the following: 1) EGFR and ALK testing in lung cancer; 2) KRAS testing in colorectal cancer; 3) BRAF testing in melanoma; and 4) HER2 testing in breast cancer. Will itemize each guideline recommendation and determine whether each pathology practice has reflexive testing protocols through self-report on the assessment. The proportion of pathology practices and exact 95% two-sided confidence intervals with reflexive-testing protocols will be calculated.
Average turnaround time of no more than 10 business days for combined EGFR and ALK results reporting in lung cancer | Up to 9 months
  The pathology practices will indicate the average number of business days between the day the tumor tissue is available and the day that all the test results are reported to the physician. Pathology practices will be considered meeting guidelines if the average is less than or equal to 10 days. The proportion of pathology practices and exact 95% two-sided confidence intervals with average turnaround time within 10 business days will be calculated.
Factors influencing heterogeneity of capacity for biomarker testing, from among modifiable testing practice-related factors, e.g. cost, complexity, technologic complexity, lack of familiarity, physician and patient demand | Up to 9 months
  For each biomarker-cancer combination being investigated, univariate and multivariate logistic regression modelling will be performed. There will be variables collected at the oncology component/subcomponent level and variables collected at the pathology practice level. The analysis will be completed at the level of the pathology practice, so characteristics of the oncology component/subcomponent will have to be adapted to that of the pathology practice: repeated for all of pathology practices used by one oncology component/subcomponent, or consolidated for pathology practices that service multiple oncology component/subcomponent. Variables used to assess heterogeneity will be (a) component/subcomponent characteristics: geography (census region), size (number of adult oncology beds), safety-net hospital, minority/underserved National Cancer Institute (NCI) Community Oncology Research Program (NCORP) component/subcomponent, academic hospital, public-ownership type.

SECONDARY OUTCOMES:
Use of genotyping or broad molecular profiling/next generation tumor sequencing for EGFR and ALK testing in lung cancer | Up to 9 months
  Will determine whether each pathology practice is using genotyping or broad molecular profiling / next-generation tumor sequencing through self reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals testing in this manner will be calculated.
Use of MMR protein expression testing by immunohistochemistry (IHC) or microsatellite instability (MSI) in colorectal cancer | Up to 9 months
  For colorectal cancer, will determine whether each pathology practice is using MMR protein expression testing by IHC or MSI through self-reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals testing in this manner will be calculated.
Capacity to test for cMET or PTEN in lung cancer | Up to 9 months
  Will determine whether each pathology practice has the capacity to test for cMET or PTEN through self-reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals with the capacity will be calculated.
Capacity to test for HRAS, AKT1, PTEN or PIK3CA in colorectal cancer | Up to 9 months
  For colorectal cancer, will determine whether each pathology practice has the capacity to test for HRAS, AKT1, PTEN or PIK3CA through self-reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals with the capacity will be calculated.
Reason for testing novel biomarkers (used for clinical care, clinical trials, or both) | Up to 9 months
  For novel biomarkers, will determine whether each pathology practice tests for novel biomarkers to be used for clinical care, clinical trials, or both through self-reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals for each time point will be calculated.
Number of days between sample availability and report availability for all biomarkers tested | Up to 9 months
  Each pathology practice will report the number of days until all biomarkers tested are completed. The average number of days across all pathology practices and 95% two-sided confidence intervals will be calculated.
Proportion of pathology practices testing for novel biomarkers using a standard reflexive testing protocol | Up to 9 months
  Will determine whether each pathology practice tests for novel biomarkers using a standard reflexive testing protocol through self-reported behavior. The proportion of pathology practices and exact 95% two-sided confidence intervals for each characteristic will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Trosman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- Center for Business Models in Healthcare, Chicago, Illinois, United States